CLINICAL TRIAL: NCT02606877
Title: Investigation of Drug-drug Interaction Between Nintedanib and Pirfenidone in Patients With IPF (an Open Label, Multiple-dose, Two Group Study)
Brief Title: A Study to Compare the Amount of Nintedanib and Pirfenidone in the Blood When Nintedanib and Pirfenidone Are Given Separately or in Combination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.229; 2015-000732-15 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

ARMS (2):
- Treatment naïve (Experimental): Treatment naïve to pirfenidone
  Interventions: Drug: nintedanib; Drug: pirfenidone
- Pirfenidone-treated (Experimental): Treatment before with pirfenidone
  Interventions: Drug: nintedanib; Drug: pirfenidone

INTERVENTIONS:
Drug: nintedanib
Drug: pirfenidone

SUMMARY:
The primary objective of this study is to investigate the effect of steady state pirfenidone on the pharmacokinetics of nintedanib and its metabolites following oral administration of 2403 mg/day pirfenidone and to investigate the effect of steady state nintedanib on the pharmacokinetics of pirfenidone at steady state following oral administration of 150 mg bid nintedanib. There will be two cohorts of patients; the first one will consist of patients not treated with pirfenidone or nintedanib, while the second one will consist of patients on pirfenidone treatment.

ELIGIBILITY:
Inclusion criteria:

Any patients diagnosed with IPF and who comply with eligibility requirements may qualify for participation in the trial.

* Written informed consent consistent with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local laws, signed prior to any study procedures being performed (including any required washout).
* Male or female patients aged >=40 years at Visit 1
* IPF diagnosis, based upon the American Thoracic Society (ATS)/European Respiratory Society(ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) 2011 guideline and chest high-resolution computed tomography (HRCT) scan.
* Force Vital Capacity (FVC) >=50% of predicted normal at Visit 1
* Diffusing capacity of the Lung for Carbon monoxide (DLCO) (corrected for Hb [visit 1]): 30%-79% predicted of normal at visit 2. (test can be performed at visits 1 or 2, or during the screening period)
* Currently treated with pirfenidone at full dose (this is only for patients going into Group 2).

Exclusion criteria:

* Alanine transaminase (ALT), Aspartate aminotransferase (AST) >1.5 fold upper limit of normal (ULN) at visit 1.
* Total bilirubin >1.5 fold ULN at visit 1.
* Underlying chronic liver disease (Child Pugh A, B, or C hepatic impairment)
* Relevant airways obstruction (i.e. pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1)/FVC <0.7 at visit 1).
* History of myocardial infarction within 6 months of visit 1 or unstable angina within 1 month of visit 1.
* Bleeding Risk:
* Known genetic predisposition to bleeding
* Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, dabigatran, heparin, hirudin, etc.) or high dose antiplatelet therapy.
* History of haemorrhagic central nervous system (CNS) event within 12 months prior to visit 1.
* History of haemoptysis or haematuria, active gastro-intestinal bleeding or ulcers and/or major injury or surgery within 3 months prior to visit 1.
* International normalised ratio (INR) >2 at visit 1.
* Prothrombin time (PT) and partial thromboplastin time (PTT) >150% of institutional ULN at visit 1.
* Planned major surgery during the trial participation, including lung transplantation, major abdominal or major intestinal surgery.
* History of thrombotic event (including stroke and transient ischemic attack) within 12 months of visit 1.
* Severe renal impairment (Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula at visit 1) or end-stage renal disease requiring dialysis.
* Treatment with n-acetylcysteine, prednisone >15 mg daily or >30 mg every 2 days OR equivalent dose of other oral corticosteroids or fluvoxamine within 2 weeks of visit 2.
* Treatment with azathioprine, cyclophosphamide, cyclosporine as well as any other investigational drug within 8 weeks of visit 2.
* Previous treatment with pirfenidone in the past three months prior to Visit 2 (Group 1 only).
* Previous treatment with nintedanib in the past 14 days prior to Visit 2.
* Permanent discontinuation of nintedanib or pirfenidone in the past due to adverse events considered drug-related.
* Known hypersensitivity to nintedanib, pirfenidone or their excipients; or to peanut or soya.
* A disease or condition which in the opinion of the investigator may interfere with testing procedures or put the patient at risk when participating in this trial.
* Alcohol or drug abuse, which in the opinion of the treating physician would interfere with treatment.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Women of childbearing potential not using highly effective methods of birth control per ICH M3, note 3, highly effective methods of birth control are defined as those, alone or in combination, that result in a low failure rate of less than 1% per year when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner. Barrier contraceptives (e.g. male condom or diaphragm) are acceptable if used in combination with spermicides (e.g. foam, gel). Contraception must be used for 28 days prior to and 3 months after nintedanib and pirfenidone administration.
* Patients not able to understand and follow study procedures including completion of diaries without help.
* Current smoker (vaping and e-cigarettes are acceptable)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (9):
- United Kingdom (9):
  - Southmead Hospital, Bristol
  - Papworth Hospital, Cambridge
  - Glenfield Hospital, Leicester
  - University College London Hospital, London
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, multiple-dose, 2-group trial in patients with idiopathic pulmonary fibrosis (IPF) to investigate the relative bioavailability of nintedanib and pirfenidone when administered alone and after coadministration.
Pre-assignment Details: Each patient group was treated according to a fixed sequence design, first with single treatment (R1, R2 respectively) followed by a combined treatment (T1, T2 respectively) which also included an up-titration period. Therefore, generating individual participant flow for each treatment group was not planned in this trial.
Groups:
- Treatment naïve: A single dose of 150 mg nintedanib (R1) was administered alone and, after pirfenidone up-titration, single dose of 150mg in combination with 801 mg tid pirfenidone (T1). Patients administered capsules orally with food.
- Pirfenidone-treated: Pirfenidone (R2) 801 mg tid was administered alone for 7 days as well as in combination with 150 mg bid nintedanib for another 7 days (T2). Patients administered capsules orally with food.
Period: Overall Study
Arm/Group | Treatment naïve | Pirfenidone-treated
Started | 20 | 17
Completed | 16 | 16
Not Completed | 4 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Non-compliance with protocol | 0 | 1
Not completed — Other than listed above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS includes all patients who received at least 1 dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment naïve | Pirfenidone-treated | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (7.8) | 68.3 (7.4) | 70.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment naïve, Area Under the Concentration-time Curve of the Nintedanib in Plasma Over the Time Interval 0 to the Last Quantifiable Data Point (AUC0-tz).
Description: AUC0-tz , area under the concentration-time curve of nintedanib in plasma over the time interval from 0 to the last quantifiable concentration. Standard error mentioned in the Method of Dispersion is actually a Geometric Standard Error.
Time Frame: Blood samples were collected at pre-dose and at 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00 and 10:00 hours post dose.
Population: Pharmacokinetic Analysis Set (PKS) - The PKS includes all patients in the treated set with at least one evaluable primary or secondary PK endpoint. (Observed cases)
Measure: Geometric Mean (Standard Error); unit: nanogram*hour/mililitre [ng*h/mL]
Groups:
- Nintedanib + Pirfenidone (T1): A single dose of 150 mg nintedanib in combination with 801 mg tid pirfenidone (T1) at day 23.
- Nintedanib (R1): A single dose of 150 mg nintedanib soft gelatin capsules was administered alone (R1) at day 1.
Arm/Group | Nintedanib + Pirfenidone (T1) | Nintedanib (R1)
Number analyzed (Participants) | 12 | 17
nanogram*hour/mililitre [ng*h/mL] | 150.31 (1.18) | 169.69 (1.15)
Statistical Analysis 1: Comparison: Nintedanib + Pirfenidone (T1) vs Nintedanib (R1); Test type: Other; ANOVA; The analysis of variance (ANOVA) model on a logarithmic scale including effects: 'subject' and 'treatment'; T1/R1 Ratio (%) = 88.58, 90% CI 2-sided [65.40 to 119.97], Standard Deviation 45.1 — To get,geometric mean ratio and Confidence Interval,least square estimates of log-transformed PK endpoint for T1 and R1 were back transformed to original scale. Standard Deviation is actually the intra-individual geometric Coefficient of Variance(%)

2. Primary Outcome: Treatment naïve, Maximum Measured Concentration of Nintedanib in Plasma After Single Dose Administration (Cmax).
Description: Cmax, maximum measured concentration of nintedanib in plasma. Standard error mentioned in the Method of Dispersion is actually a Geometric Standard Error.
Time Frame: Blood samples were collected at pre-dose and at 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00 and 10:00 hours post dose.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanogram/mililitre [ng/mL]
Arm/Group | Nintedanib + Pirfenidone (T1) | Nintedanib (R1)
Number analyzed (Participants) | 12 | 17
nanogram/mililitre [ng/mL] | 23.04 (1.23) | 28.58 (1.19)
Statistical Analysis 1: Comparison: Nintedanib + Pirfenidone (T1) vs Nintedanib (R1); Test type: Other; ANOVA; The analysis of variance (ANOVA) model on a logarithmic scale including effects: 'subject' and 'treatment'; T1/R1 Ratio (%) = 80.63, 90% CI 2-sided [51.27 to 126.79], Standard Deviation 74.6 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Pirfenidone-treated, Area Under the Concentration-time Curve of Pirfenidone in Plasma Over a Dosing Interval at Steady State (AUCτ,ss)
Description: AUCτ,ss, area under the concentration-time curve of pirfenidone in plasma over a dosing interval at steady state. Standard error mentioned in the Method of Dispersion is actually a Geometric Standard Error.
Time Frame: Blood samples were collected at pre-dose and at 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00 and 10:00 hours post dose.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanogram*hour/mililitre [ng*h/mL]
Groups:
- Pirfenidone+Nintedanib (T2): Pirfenidone 801 mg tid was administered in combination with 150 mg bid nintedanib for 7 days.
- Pirfenidone (R2): Pirfenidone 801 mg tid was administered alone for 7 days.
Arm/Group | Pirfenidone+Nintedanib (T2) | Pirfenidone (R2)
Number analyzed (Participants) | 13 | 15
nanogram*hour/mililitre [ng*h/mL] | 39040.84 (1.07) | 40178.46 (1.07)
Statistical Analysis 1: Comparison: Pirfenidone+Nintedanib (T2) vs Pirfenidone (R2); Test type: Other; ANOVA; The analysis of variance (ANOVA) model on a logarithmic scale including effects: 'subject' and 'treatment'; T2/R2 Ratio (%) = 97.17, 90% CI 2-sided [87.84 to 107.48], Standard Deviation 14.1 — To get,geometric mean ratio and Confidence Interval,least square estimates of log-transformed PK endpoint for T2 and R2 were back transformed to original scale. Standard Deviation is actually the intra-individual geometric Coefficient of Variance(%)

4. Primary Outcome: Pirfenidone-treated, Maximum Measured Concentration of Pirfenidone in Plasma at Steady State (Cmax,ss)
Description: Cmax,ss, maximum measured concentration of pirfenidone in plasma at steady state. Standard error mentioned in the Method of Dispersion is actually a Geometric Standard Error.
Time Frame: Blood samples were collected at pre-dose and at 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00 and 10:00 hours post dose.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanogram/mililitre [ng/mL]
Arm/Group | Pirfenidone+Nintedanib (T2) | Pirfenidone (R2)
Number analyzed (Participants) | 13 | 15
nanogram/mililitre [ng/mL] | 10537.26 (1.08) | 10591.08 (1.08)
Statistical Analysis 1: Comparison: Pirfenidone+Nintedanib (T2) vs Pirfenidone (R2); Test type: Other; ANOVA; The analysis of variance (ANOVA) model on a logarithmic scale including effects: 'subject' and 'treatment'; T2/R2 Ratio (%) = 99.49, 90% CI 2-sided [87.94 to 112.56], Standard Deviation 17.4 — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Treatment naïve, Area Under the Concentration-time Curve of Nintedanib in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of nintedanib in plasma over the time interval from 0 extrapolated to infinity. Standard error mentioned in the Method of Dispersion is actually a Geometric Standard Error.
Time Frame: Blood samples were collected at pre-dose and at 0:30, 1:00, 2:00, 3:00, 4:00, 6:00, 8:00 and 10:00 hours post dose.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: nanogram*hour/mililitre [ng*h/mL]
Arm/Group | Nintedanib + Pirfenidone (T1) | Nintedanib (R1)
Number analyzed (Participants) | 12 | 17
nanogram*hour/mililitre [ng*h/mL] | 175.04 (1.18) | 195.59 (1.15)
Statistical Analysis 1: Comparison: Nintedanib + Pirfenidone (T1) vs Nintedanib (R1); Test type: Other; ANOVA; The analysis of variance (ANOVA) model on a logarithmic scale including effects: 'subject' and 'treatment'; T1/R1 Ratio (%) = 89.49, 90% CI 2-sided [66.33 to 120.73], Standard Deviation 44.3 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after last drug administration, up to 6 weeks.
Description: The assessment of safety was a further objective of the trial. Due to the study design, there was a great difference in duration of treatment reference (R) and treatment (T) within each patient group and a long residual effect period of the first treatment that overlapped with the second treatment. Thus the study design did not allow for a reliable comparison of treatment R and T within each patient group regarding safety and the trial team decided to provide the safety assessment only overall.
Arm/Group | Treatment naïve | Pirfenidone-treated
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 13/20 | 15/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment naïve (N=20) | Pirfenidone-treated (N=17)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall mass (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 3
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Fatigue (General disorders) | 4 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Blood pressure increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Ageusia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 5 | 0
Presyncope (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT02606877/SAP_000.pdf
  • Study Protocol (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT02606877/Prot_001.pdf